CLINICAL TRIAL: NCT05279365
Title: PROSPECTIVE OPEN LABEL CLINICAL TRIAL TO ADMINISTER A BOOSTER DOSE OF PFIZER/BIONTECH OR MODERNA COVID-19 VACCINE IN HIGH-RISK INDIVIDUALS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DHR Health Institute for Research and Development (Other)
Responsible Party: Principal Investigator, Sohail Rao, President & Chief Executive Officer, DHR Health Institute for Research and Development
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1789039
Record Dates: First submitted 2022-03-14; First posted 2022-03-15 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: SARS CoV 2 Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of Booster Dose (Experimental): study participant will receive either 30ug in 0.3 ml of Pfizer/BioNTech (BNT162b2) or 0.25 ml of Moderna vaccine administered intramuscularly.
  Interventions: Biological: Pfizer/BioNTech (BNT162b2); Biological: Moderna

INTERVENTIONS:
Biological: Pfizer/BioNTech (BNT162b2) — participants will receive a booster dose (1st booster or 2nd booster) of vaccine
Biological: Moderna — participants will receive a booster dose (1st booster or 2nd booster) of vaccine

SUMMARY:
The recent rise in infections with the Omicron variant of the SARS-CoV-2 is alarming. Equally disconcerting is the fact that individuals who were previously vaccinated (< 6 months) and have co-morbidities that are considered high risk, are getting re-infected...a process referred to as "breakthrough". There is some evidence that in these high risk individuals, the gradual decrease in immunity against the virus as depicted by a drop in anti-SARS-CoV-2 antibodies, is responsible (partially or wholly) for this reinfection. In this study, we intend to give a booster does Pfizer/BioNTech and/or Moderna and ascertain the levels of antibodies at various times pre and post vaccination. The incidence of infection with SARS-CoV-2 after booster vaccination will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and over that have been fully vaccinated (2 doses) with the Pfizer/BioNTech COVID-19 vaccine (BNT162b2) and with the 1st booster at least 90 days prior to the 2nd booster
* Healthcare workers employed by and/or affiliated with DHR Health, Renaissance Medical Foundation, DHR Partners, Starr County Memorial Hospital
* Any adult with any of the following risk factors for severe COVID-19 disease progression (as outlined by the CDC)

Exclusion Criteria:

* Previous history of allergic reaction to vaccination
* less than or equal to 3 months from last booster dose of vaccine
* active SARS-COV-2 infection
* less than or equal to 21 days of full recovery from SARS-CoV-2 infection
* less than or equal to 14 days of any vaccination
* vaccinated with any other available COVID-19 vaccine other than Pfizer/BioNTech or Moderna
* Healthcare workers not employed by and/or affiliated with DHR Health, Renaissance Medical Foundation, Star County Memorial Hospital or non DHR Partners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants infected with SARS-CoV-2 after booster Dose | 24 months
  Determine effectiveness of booster dose in the prevention of SARS-CoV-2 Infection by assessing if subjects remain free from infections with SARS-CoV-2 after receiving booster dose.
Levels of anti-SARS-CoV-2 IgG antibody titers after booster | 24 months
  Determine the anti-SARS-CoV-2 IgG antibody titers using a semi quantitative method at various time points (Baseline/Day 0, Day 14, Week 12 and Week 24 after booster) to assess for sustained levels of relatively high titers of anti-SARS-CoV-2 IgG in the blood of the subjects

SECONDARY OUTCOMES:
Measure rate of decline of immune responses | 24 months
  Determine the rate of decline of immune responses in various cohort of recipients with similar co-morbidities by conducting cohort analysis
Identify differences in immune responses based on comorbidity status | 24 months
  Identify differences in immune responses based on comorbidity status (e.g., Immune response in recipients with metabolic diseases vs. patients with immunosuppression) by using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Rao, MD,MA,DPhil, Principal Investigator — DHR Health Institute for Research and Development
Locations (4):
- United States (4):
  - Brownsville Independent School District, Brownsville, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - Edinburg CISD School Based Health Center, Edinburg, Texas
  - Starr County Memorial Hospital, Rio Grande City, Texas

IPD SHARING:
Plan to Share IPD: No